CLINICAL TRIAL: NCT03427619
Title: A Phase 2, Multicenter, Open Label Study to Evaluate the Efficacy and Safety of OK-432 Immunotherapy in Individuals With Lymphatic Malformations
Brief Title: OK432 (Picibanil) in the Treatment of Lymphatic Malformations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard JH Smith (Other)
Responsible Party: Sponsor-Investigator, Richard JH Smith, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201107741
Record Dates: First submitted 2018-01-10; First posted 2018-02-09 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Lymphatic Malformations
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Picibanil

STUDY DESIGN:
Intervention Model Description: All eligible participants receive the actual drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OK432 (Picibanil) (Experimental): There is no control in this study. All participants will receive the actual drug -OK432. With each injection they may receive 0.01 to 0.05mg/mL 6-12 weeks apart up to 4 injections total.
  Interventions: Drug: OK432

INTERVENTIONS:
Drug: OK432 — OK432 will be injected at dosage of 0.01 to 0.05 mg/mL 6-12 weeks apart up to 4 injections total.
  Other Names: Picibanil

SUMMARY:
Standard of care for Lymphatic Malformations has been surgical excision. We have been using OK432/Picibanil (generously supplied by Chugai Pharmaceuticals in Japan) since 1992 with great success for macrocystic disease.

The objective of the study was to provide OK-432 immunotherapy to subjects with macrocystic or mixed (> 50% macrocystic) lymphatic malformations (LMs) and investigate the efficacy and safety of OK 432 as a treatment option in subjects with LMs.

DETAILED DESCRIPTION:
Lymphatic malformations are uncommon tumors that represent localized malformations in the development of the lymphatic system. They typically present in children under 2 years of age and in almost 50% of the cases, are diagnosed at birth. There is neither a racial nor a sexual tendency. The malformations can occur anywhere on the body, but typically they are in the head/neck area.

Morbidity can be significant. Besides the obvious cosmetic deformity caused by these tumors, there is risk of infection and airway compromise and even obstruction. However, effective therapeutic options are limited. Small lesions can be observed, although spontaneous resolution is unlikely. For larger lesions, surgery has been the traditional form of therapy. In the head and neck, in particular, lymphangiomas typically wrap themselves around major neurovascular structures, making total excision removal difficult, if not impossible, and thus the likelihood of recurrence is quite high. Because of these surgical limitations, alternate therapies have been considered; including cryotherapy, diathermy, and chemical sclerotherapy.

The investigators experience with using the drug for macrocystic disease(large cysts) since 1992 in the United States has been very promising compared to traditional surgery. Recurrence rate to date, has been very minimal as well. (<2%)

After the conclusion of the Phase 2 randomized study, all new subjects who presented with an LM and were eligible for treatment were treated under an open-label protocol for continued access to OK-432. This multicenter, open label study enrolled subjects between September 2005 and November 2017.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to receive OK432 immunotherapy

* Patients must be ages 6 months to 17 years
* Patients must have a macrocystic Lymphatic Malformation
* Patients may have had surgical treatment for their Lymphatic Malformation
* Patients must have an imaging study to confirm the diagnosis of a macrocystic or mixed Lymphatic Malformation An MRI is preferred over a CT scan (an ultrasound may be used between injections if warranted, however an MRI or CT should be done pre and post treatment)

Exclusion Criteria:

* Penicillin allergy
* Women who are pregnant or nursing
* Patients who present with a temperature of 100.5 degrees F or greater
* Patients with mixed hemangioma-lymphangioma lesions
* Patients with a history OR a family history of rheumatic heart disease or post-streptococcal glomerulonephritis
* Patients with hemodynamic instability and respiratory failure
* Patients with a history OR a family history of obsessive-compulsive, tic disorders, or PANDA (pediatric autoimmune neuro-psychiatric disorder associated with streptococcal infections)
* Patients who demonstrate abnormalities in the history, physical examination or laboratory analysis which may indicate significant hepatic, hematologic, or renal disease
* Patients who are not in "good general health" (including patients with congenital disorders, chronic diseases, immunologic dysfunction, transplant recipients)

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2005-10-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard JH Smith, MD, Principal Investigator — University of Iowa
Locations (14):
- United States (14):
  - Rady Children's Hospital & Health Center San Diego, San Diego, California
  - The Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Richard Smith, MD, Iowa City, Iowa
  - Spectrum Health-SHMG Ear, Nose, & Throat, Grand Rapids, Michigan
  - Children's Hospitals & Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - SUNY Health Science Center, Syracuse, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Vanderbilt University Hospital, Nashville, Tennessee
  - Children's ENT of Houston, Houston, Texas
  - Children's Hospital of the Kings Daughter, Norfolk, Virginia
  - University of Wisconsin Hospital & Clinic, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 14 centers across the United States between September 2005 and November 2017.
Pre-assignment Details: After informed consent, subjects who met all eligibility criteria were enrolled into the study. Study completion data was analyzed retrospectively for subjects with observed, non-missing data.
  Results presented in this report were based on a retrospective analysis of source-verified data and therefore only non-missing data is presented. Therefore there are differences in the number of subjects for different analyses.
Groups:
- OK-432: OK 432 is a lyophilized biological preparation for injection containing nonviable cells of Streptococcus pyogenes (A group, type 3) Su strain treated with benzylpenicillin.
  OK-432 was administered intracystically at a concentration of 0.01 to 0.05 mg/mL. A 4-dose injection series of OK-432 was planned for all subjects. All injections were spaced approximately 6 to 12 weeks apart
Period: Overall Study
Arm/Group | OK-432
Started | 275
Safety Population | 275
Modified Intention to Treat Population | 143
Completed | 209
Not Completed | 66
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 5
Not completed — Administrative | 4
Not completed — Other | 2
Not completed — Unknown or Missing Completion Status | 48

BASELINE CHARACTERISTICS:
Population: The Safety Population included all enrolled subjects that have been treated with at least one injection of OK-432. Results were based on a retrospective analysis of source-verified data and only non-missing data is presented. Therefore there are differences in the number of subjects for different analyses.
Arm/Group | OK-432
Number analyzed (Participants) | 275
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic information for age was available for 273 subjects. Missing for 2 subjects.
  years
    number analyzed (Participants) | 273
    (all) | 5.481 (6.6382)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic information for gender was available for 274 subjects. Missing for 1 subject.
  Participants
    number analyzed (Participants) | 274
    Female | 151
    Male | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Demographic data on race/ethnicity was available for 266 subjects. Data was missing for 9 subjects. Please note that participants could report more than one Race/Ethnicity.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 266
    Hispanic or Latino | 36
    American Indian or Alaska Native: number analyzed (Participants) | 266
    American Indian or Alaska Native | 2
    White: number analyzed (Participants) | 266
    White | 191
    Black or African American: number analyzed (Participants) | 266
    Black or African American | 29
    Asian: number analyzed (Participants) | 266
    Asian | 10
    Other: number analyzed (Participants) | 266
    Other | 7
Region of Enrollment [Number; unit: participants]
  United States | 275

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success at 1 to 6 Months Post-Therapy as Assessed by Imaging
Description: Clinical success was defined as having either a complete (90% 100%) or substantial (60% 89%) reduction in lymphatic malformation (LM) volume after treatment. Response was determined using post treatment imaging studies at approximately 1 to 6 months after completion of treatment
Time Frame: 1 to 6 Months Post-Therapy
Population: The modified Intent to Treat (mITT) Population includes all enrolled subjects treated with at least one injection of OK 432 who either have post-therapy imaging assessment data or at least one investigator assessment of overall response throughout the study (N = 148). The efficacy data were presented as observed for subjects with non-missing data in the mITT Population (N = 78).
Measure: Count of Participants; unit: Participants
Arm/Group | OK-432
Number analyzed (Participants) | 78
Participants | 57

2. Secondary Outcome: Number of Participants With Clinical Response 1 to 6 Months Post-Therapy as Assessed by Imaging
Description: Number of participants who demonstrated a complete (90%-100% reduction in LM volume), substantial (60%-89% reduction in LM volume), intermediate (20%-59% reduction in LM volume), or no (< 20% reduction in LM volume) response 1 to 6 months post-therapy as assessed by imaging
Time Frame: 1 to 6 Months Post-Therapy
Population: The mITT includes all enrolled subjects treated with at least one injection of OK 432 who either have post-therapy imaging assessment data or at least one investigator assessment of overall response throughout the study (N = 148). The efficacy data were presented as observed for subjects with non-missing data in the mITT Population (N = 78).
Measure: Count of Participants; unit: Participants
Arm/Group | OK-432
Number analyzed (Participants) | 78
Participants
  Number of subjects who achieved a complete response | 43
  Number of subjects who achieved a substantial response | 14
  Number of subjects who achieved an intermediate response | 5
  Number of subjects who achieved no response | 16

3. Secondary Outcome: Number of Participants With Investigator-Evaluated Overall Response
Description: Investigator evaluated post-therapy clinical response based on physical exam and/or ultrasound was categorized as "Clinical Improvement" or "No Change" in the size of the cyst.
Time Frame: 1 to 6 Months Post-Therapy
Population: The mITT Population includes all enrolled subjects treated with at least one injection of OK 432 who either have post-therapy imaging assessment data or at least one investigator assessment of overall response throughout the study (N = 148). The investigator assessed response data were presented as observed for subjects with non-missing data in the mITT Population (N = 98).
Measure: Count of Participants; unit: Participants
Arm/Group | OK-432
Number analyzed (Participants) | 98
Participants | 80

4. Secondary Outcome: Change From Baseline in Lesion Volume
Description: Percent change from baseline in lesion volume - pre-therapy to post therapy assessed by imaging.
Time Frame: Baseline and 1 to 6 Months Post-Therapy
Population: The mITT includes all enrolled subjects treated with at least one injection of OK 432 who either have post-therapy imaging assessment data or at least one investigator assessment of overall response throughout the study (N = 148). The efficacy data were presented as observed for subjects with non-missing data in the mITT Population (N = 76).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | OK-432
Number analyzed (Participants) | 76
percent change | -44.92 (110.561)

ADVERSE EVENTS:
Time Frame: Nonserious AEs (Subject Diary): Up to 14 days after each injection Treatment Emergent SAEs: Day 1 to 35 days after last injection All Cause Mortality: Day 1 to study completion ie, 2 years after treatment completion (All-Cause Mortality) Note: Results presented were based on a retrospective analysis of source-verified data and therefore only non-missing data is presented. Therefore there are differences in the number of subjects for different analyses.
Description: In this study, "serious adverse event" (SAE) was defined as any deviation from expected response to OK-432 immunotherapy. Treatment emergent SAE (TESAE) was defined as any SAE occurring or worsening on or after the first dose of study drug and within 35 days after the last dose of study drug.
  Other AEs were collected via Subject Diaries were presented as observed for subjects who provided diary data. Therefore the participants at risk for Other AEs (N = 114) is less than for SAEs (N = 275)
Arm/Group | OK-432
All-Cause Mortality (participants affected / at risk) | 0/275
Serious Adverse Events (participants affected / at risk) | 11/275
Other Adverse Events (participants affected / at risk) | 112/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OK-432 (N=275)
Pyrexia (General disorders) | 5
Injection site swelling (General disorders) | 2
Swelling (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Odynophagia (Gastrointestinal disorders) | 1
Furuncle (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Bradycardia (Cardiac disorders) | 1
Milk allergy (Immune system disorders) | 1
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1
Febrile convulsion (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OK-432 (N=114)
Swelling (General disorders) | 112
Pain (General disorders) | 112
Redness (General disorders) | 110
Fever (General disorders) | 72
Fatigue (General disorders) | 66
Decreased appetite (General disorders) | 63
Nausea/vomiting (General disorders) | 35
Headache (General disorders) | 32
Chills (General disorders) | 21
Joint pain (General disorders) | 18
Rash (General disorders) | 7

LIMITATIONS AND CAVEATS:
Results are based on a retrospective analysis of source-verified data that include subjects enrolled in the open label study. This study was conducted to provide patients with continued access to OK-432 on a compassionate use basis. Response data were not well documented for everyone. Subjects with missing data included those who were lost to follow up, had incomplete or missing CRFs or imaging studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03427619/Prot_SAP_000.pdf